CLINICAL TRIAL: NCT07083648
Title: Magnetic Resonance Imaging-guided Online Adaptive Radiotherapy Using a Dedicated MR-simulator and a Cone Beam CT Based Treatment Delivery for Stereotactic Body Radiation Therapy of Pelvic Lymph Node Metastases (MACULA-Trial)
Brief Title: Magnetic Resonance Imaging-guided Online Adaptive Radiotherapy of Pelvic Lymph Node Metastases
Acronym: MACULA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAO-24-017
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pelvic and Para-aortic Lymph Node Metastases
Keywords: pelvic; lymph node; para-aortic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided online adaptive RT using a dedicated MR-simulator and cone-beam CT (CBCT)-based treatment (Experimental)
  Interventions: Radiation: Magnetic resonance Imaging-guided online adaptive radiotherapy

INTERVENTIONS:
Radiation: Magnetic resonance Imaging-guided online adaptive radiotherapy — On each day of treatment, a new MRI scan in the treatment position will be acquired using the dedicated MR simulator, co-registered with the original one. The original target and organ at risk (OAR) contours will be propagated to the new image set using rigid and deformable image registration. The contours will be adapted to changes detected with MRI of the day. The original SBRT treatment plan will be adapted to the changed and hence adapted anatomy of targets and OARs by plan optimization. Dose calculation will be performed on the newly generated synthetic CT (preferred) or, if there is a contra-indication for synthetic CT, on the original image.

SUMMARY:
In this study, the investigators want to investigate whether online-adapted radiotherapy using a special magnetic resonance imaging (MRI) simulator and computed tomography (CT)-guided radiation therapy, is feasible and offers advantages for the treatment of pelvic lymph node metastases.

DETAILED DESCRIPTION:
MR-guided online adaptive radiotherapy has been implemented recently using MR-linac technology, where MR-imaging is combined with linac technology in hybrid systems. These systems offer MR imaging for online adaptive radiotherapy (RT) within the treatment room and with the patient in treatment position. Despite results regarding technical and clinical feasibility being promising, the high costs of MR-linacs systems and the high demands for staffing resources of MR-linacs are limiting a boarder implementation of this technology. At the Department of Radiation Oncology, University Hospital Zurich, MRI-simulations for RT planning using a dedicated scanner have been performed since 2023. The investigators have developed and implemented an MRI-only RT planning workflow followed by RT delivered at a CBCT-guided, conventional linac. The aim to expand the MRI-only workflow to online adaptive RT. This study will investigate the feasibility of MRI-guided, online adaptive SBRT for pelvic and para-aortic lymph node metastases using a dedicated MR simulator and treatment delivery using conventional CBCT-linac technology.

ELIGIBILITY:
Inclusion Criteria:

* Intra-pelvic and para-aortic lymph node metastases from a histologically confirmed malignancy;
* Indication for SBRT based on a multidisciplinary tumor board recommendation and / or clinical practice guideline;
* Intra-pelvic and para-aortic lymph node metastases confirmed by imaging and amenable for SBRT

Exclusion Criteria:

* Large body size that would not fit the MRI-simulator bore;
* Contraindications for MRI including but not limited to

  * electronic devices such as pacemakers, defibrillators, deep brain stimulators, cochlear implants that are labeled as MR unsafe. Electronic devices labeled as MR safe or MR conditional are not a contraindication;
  * metallic foreign body in the eye or aneurysm clips in the brain;
  * severe claustrophobia;
  * hip prosthesis that are labeled as MR unsafe;
* More than 5 pelvic lymph node metastasis
* Previous radiation therapy directly overlapping with SBRT in this study and leading to exceeding tolerance of OARs;
* History of Crohn's disease, ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Rate of successfully delivered fractions | during treatment, 1-2 weeks
  Feasibility is measured as a successful delivery of an MRI-adapted plan using CBCT image-guidance in another room in 90% of the SBRT fractions.

SECONDARY OUTCOMES:
Average improvement of coverage of planning target volume | During treatment, 1-2 weeks
  Dosimetric advantage is defined as >5% improvement in coverage of the planning target volume (PTV) or >5% better sparing of one of the organs at risk (bowel, sigma , rectum, bladder).
Adverse Events | during SBRT, 3 months and 24 months of follow-up
  Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich University Hospital, Department of Radiation Oncology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided